CLINICAL TRIAL: NCT00699764
Title: Safety of SmithKline Beecham Biologicals' Herpes Simplex Candidate Vaccine (gD2t) With MPL & Its Efficacy to Prevent Genital Herpes Disease in HSV Positive or Negative Consorts of Subjects With Genital Herpes Disease
Brief Title: Safety of a Herpes Simplex Candidate Vaccine (gD2t) With MPL and Its Efficacy to Prevent Genital Herpes Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 208141/017
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Herpes Simplex
Keywords: Herpes simplex candidate vaccine; Herpes simplex
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental)
  Interventions: Biological: Herpes simplex candidate vaccine- adjuvanted GSK208141
- Group B (Placebo Comparator)
  Interventions: Biological: Placebo injection

INTERVENTIONS:
Biological: Herpes simplex candidate vaccine- adjuvanted GSK208141 — Intramuscular injection, 3 doses
  Arms: Group A
Biological: Placebo injection — Intramuscular injection, 3 doses
  Other Names: Herpes simplex candidate vaccine- adjuvanted GSK208141
  Arms: Group B

SUMMARY:
The purpose of the study is to evaluate the safety of Herpes Simplex candidate vaccine (gD2t) with adjuvant and its efficacy to prevent genital herpes disease in HSV positive or negative consorts of subjects with genital herpes disease.

DETAILED DESCRIPTION:
This study was monitored by a Data Safety Monitoring Board At the time of conduct of this study, the sponsor GlaxoSmithKline was known by its former name SmithKline Beecham

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 45 years of age at the time of first vaccination
* Written informed consent
* Females of childbearing potential must have a negative pregnancy test at enrollment and be using an accepted method of birth control
* The volunteers must have a regular sexual partner with genital herpes disease confirmed by medical history

Exclusion Criteria:

* Any previous history of or current clinical signs or symptoms of genital herpes disease.
* Any previous vaccination against herpes simplex.
* Any previous administration of MPL.
* History of herpetic keratitis.
* History of erythema multiforme.
* Female subjects who are pregnant, lactating or planning a pregnancy before one month after the last vaccine dose.
* Patient is immuno-compromised or is receiving immuno-modifying therapy of any kind. Topical corticoid therapy is allowed.
* HIV positive at the time of enrollment
* Clinical signs of acute or febrile illness at the time of entry into the study.
* Any continuous suppressive antiviral oral therapy within the 6 months prior to entry.
* Any administration of immunoglobulins during the vaccination course or within one month prior to the first vaccination.
* Any vaccine administration less than one week before or after a study vaccination.
* Previous known hypersensitivity to vaccination or to any component of the vaccine.
* Simultaneous participation in any other clinical trial of an investigational compound.
* Recent history of alcoholism or drug abuse
* Recent clinical history or evidence of significant hepatic disease
* Recent clinical history or evidence of renal dysfunction
* Life-threatening or serious cardiac (NYHA grades III-IV), gastrointestinal, haematological or immunological disorder which, in the opinion of the investigator, would preclude entry into the study.
* Inability or unwillingness to comply with the protocol or not expected to complete the study period

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2491 (Actual)
Dates: Start 1996-03; Primary Completion 1999-10 (Actual); Study Completion 1999-10 (Actual)

PRIMARY OUTCOMES:
To compare between herpes simplex vaccine (gD2t with adjuvant) and placebo the general safety of the vaccine by recording all the unsolicited adverse experiences | During the 7 month vaccination period
To evaluate the protective efficacy of gD2t with adjuvant to prevent acquisition of genital herpes disease in healthy female adults who are HSV seronegative or HSV seropositive at baseline | Survival analysis beginning at Month 0

SECONDARY OUTCOMES:
To evaluate the protective efficacy of gD2t with adjuvant vaccine to prevent acquisition of genital herpes disease in healthy female adults who are HSV seronegative at baseline | Survival analysis beginning at Month 0
To evaluate the protective efficacy of the gD2t with adjuvant vaccine to prevent acquisition of genital herpes disease in healthy male and female adults who are HSV seronegative or HSV-1 seropositive at baseline | Survival analysis beginning at Month 0
To evaluate the protective efficacy of the gD2t with adjuvant vaccine to prevent acquisition of genital herpes disease in healthy female adults who are HSV seronegative or HSV-1 seropositive at baseline | After 3 doses of vaccine (between months 7 and 19)
To evaluate the protective efficacy of the gD2t with adjuvant vaccine to prevent symptoms of genital herpes disease in healthy female adults who are HSV seronegative at baseline | Survival analysis beginning at Month 0
To evaluate the protective efficacy of gD2t with adjuvant vaccine to prevent HSV infection in healthy female adults who are HSV seronegative or HSV-1 seropositive at baseline
To evaluate the protective efficacy of gD2t with adjuvant vaccine to prevent HSV infection in healthy female adults who are HSV seronegative at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Stanberry LR, Spruance SL, Cunningham AL, Bernstein DI, Mindel A, Sacks S, Tyring S, Aoki FY, Slaoui M, Denis M, Vandepapeliere P, Dubin G; GlaxoSmithKline Herpes Vaccine Efficacy Study Group. Glycoprotein-D-adjuvant vaccine to prevent genital herpes. N Engl J Med. 2002 Nov 21;347(21):1652-61. doi: 10.1056/NEJMoa011915. PMID 12444179
- [Background] Tavares F, Cheuvart B, Heineman T, Arellano F, Dubin G. Meta-analysis of pregnancy outcomes in pooled randomized trials on a prophylactic adjuvanted glycoprotein D subunit herpes simplex virus vaccine. Vaccine. 2013 Mar 25;31(13):1759-64. doi: 10.1016/j.vaccine.2013.01.002. Epub 2013 Jan 10. PMID 23313657
- [Background] Verstraeten T, Descamps D, David MP, Zahaf T, Hardt K, Izurieta P, Dubin G, Breuer T. Analysis of adverse events of potential autoimmune aetiology in a large integrated safety database of AS04 adjuvanted vaccines. Vaccine. 2008 Dec 2;26(51):6630-8. doi: 10.1016/j.vaccine.2008.09.049. PMID 18845199
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 208141/017 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 208141/017 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 208141/017 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 208141/017 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 208141/017 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 208141/017 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register